CLINICAL TRIAL: NCT06516653
Title: Postmarket Surveillance, Prospective, Multicenter, Randomized, Controlled Study Evaluating the Performance of VasQ for Its Intended Use.
Brief Title: Post Market Study for VasQ, an External Support Implant for Arteriovenous Fistula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laminate Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CD0261
Record Dates: First submitted 2024-07-16; First posted 2024-07-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- End to side fistula supported with VasQ (Experimental): Patients receiving an end to side arteriovenous fistula, supported by VasQ, for fistula access
  Interventions: Device: VasQ; Procedure: Arteriovenous fistula creation for dialysis vascular access
- Standard of care end to side fistula (Active Comparator): Patients receiving an end to side arteriovenous fistula, for fistula access
  Interventions: Procedure: Arteriovenous fistula creation for dialysis vascular access

INTERVENTIONS:
Device: VasQ — External support implant for the arteriovenous fistula
  Arms: End to side fistula supported with VasQ
Procedure: Arteriovenous fistula creation for dialysis vascular access — End to side fistula creation in the arm for dialysis vascular access

SUMMARY:
VasQ is an external support implant for arteriovenous fistulas created for dialysis access.

This is a postmarket surveillance, prospective, multi-center, randomized, controlled, open label trial enrolling 300 patients randomized into two study arms:

* Treatment arm: End to side fistula supported with VasQ
* Control: Standard of care end to side fistula

DETAILED DESCRIPTION:
Structure

This is a postmarket surveillance, prospective, multi-center, randomized, controlled, open label trial enrolling 300 patients randomized into two study arms:

* Treatment arm: End to side fistula supported with VasQ
* Control: Standard of care end to side fistula

Duration The primary endpoint is defined at 6 month post index procedure of fistula creation. Patients will be further followed up to 12 months post index procedure.

Main study question What is the magnitude of benefit of the VasQ device with regard to time to achieving a clinically functional AVF as compared to a comparable contemporary standard of care cohort?

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are candidates for the creation of a new radiocephalic or brachiocephalic end-to-side surgical AV fistula for dialysis access (per VasQ IFU and investigator clinical judgment) and consent to take part in the study.
2. Male and non-pregnant female participants.
3. Age 18-80 years
4. Patients willing and able (physically and geographically) to attend follow up visits over a period of 12 months.

Exclusion Criteria:

1. Index procedure being a revision surgery of an existing fistula.
2. Significantly stenotic target vein on the side of surgery (≥50%) as diagnosed on preoperative ultrasound. (Scan should include the full length of the expected fistula outflow, starting at the planned anastomosis site)
3. Unusual anatomy or vessel dimensions (observed on pre-operative ultrasound or intraoperatively) and which preclude adequate fit of the VasQ.
4. Known central venous stenosis or obstruction on the side of surgery.
5. Pre-existing stents or stent grafts in the access circuit.
6. Planned subsequent fistula superficialization procedure.
7. Known coagulation disorder.
8. Known allergy to nitinol.
9. Expected kidney transplant within 12 months of enrollment.
10. Inability to give consent and/or comply with the study follow up schedule.
11. Insufficient or borderline life expectancy to allow for completion of study procedures and follow-up (12 Months).
12. Participation in another interventional study that in the judgment of the investigator could confound study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Fistula functional success | 6 months
  The time, in days, to the first day of a 28-day period in which the study fistula was able to be cannulated with two dialysis needles for at least 75% of dialysis sessions to achieve the prescribed dialysis

OTHER OUTCOMES:
Safety - vascular access related complications | 1 year
  Comparable rate of access related complications (including major reintervention and cannulation related complications)

CONTACTS AND LOCATIONS:
Overall Officials: John F Lucas III, MD, FACS, FSVS, Principal Investigator — Greenwood Leflore Hospital
Locations (7):
- United States (7):
  - Fresenius Vascular Care Long Beach, Long Beach, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Greenwood Leflore Hospital, Greenwood, Mississippi
  - Azura Surgery Center Las Vegas, Las Vegas, Nevada
  - Fresenius Vascular Care Columbia, Columbia, South Carolina
  - Fairlawn Surgery Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No